CLINICAL TRIAL: NCT06182501
Title: Interference by Activated Protein C Resistance in the Determination of Protein S Activity
Acronym: PS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8674
Record Dates: First submitted 2022-09-06; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Resistance to Activated Protein C in the Determination of Protein S Activity
Keywords: protein C; protein S; activated protein C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protein S is an anticoagulant protein and a cofactor of protein C. It is recommended to explore it first by a functional (chronometric) technique by assessing its cofactor activity of activated protein C. Existing tests measure the prolongation of a coagulation time. These tests are all dependent on factor V, but some patients have mutations in factor V (including V Leiden) that make them resistant to activated protein C activity. It is suspected that these mutations lead to underestimations of protein S activity by chronometric technique.

ELIGIBILITY:
Inclusion criteria:

* Patient of legal age (≥ 18 years)
* Patient for whom a sample has been sent to the HUS Hematology Laboratory for measurement of protein S activity between 28/12/2009 and 29/12/2020
* Patient who does not object to the reuse of his/her medical data for scientific research purposes.

Exclusion criteria:

* Minor patient
* Patient with incomplete data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) for whom a sample has been sent to the HUS Hematology Laboratory for measurement of protein S activity between 28/12/2009 and 29/12/2020
Sampling Method: Non-Probability Sample
Enrollment: 9470 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Functional test protein C resistance | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - CHU de Strasbourg - France, Strasbourg, France